CLINICAL TRIAL: NCT01459679
Title: Multi-Center, Randomized, Controlled Evaluation of the Safety & Efficacy of the KXL System With VibeX (Riboflavin Ophthalmic Solution) for Corneal Collagen Cross-Linking in Eyes With Keratoconus or Corneal Ectasia After Refractive Surgery
Brief Title: Safety & Efficacy of Corneal Collagen Cross-Linking in Eyes With Keratoconus or Corneal Ectasia After Refractive Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: American-European Congress of Ophthalmic Surgery (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACOS-KXL-001
Record Dates: First submitted 2011-09-19; First posted 2011-10-26 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-06

CONDITIONS: Keratoconus; Corneal Ectasia
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- VibeX Treatment Group A (Active Comparator): Corneal collagen cross-linking using riboflavin ophthalmic solution and ultraviolet-A (UVA) light for 8 minutes
  Interventions: Device: KXL System (15 mW/cm2); Drug: riboflavin ophthalmic solution
- VibeX Treatment Group B (Active Comparator): Corneal collagen cross-linking using riboflavin ophthalmic solution and ultraviolet-A (UVA) light for 4 minutes
  Interventions: Device: KXL System (30 mW/cm2); Drug: riboflavin ophthalmic solution
- VibeX Treatment Group C (Active Comparator): Corneal collagen cross-linking using riboflavin ophthalmic solution and ultraviolet-A (UVA) light for 2 minutes and 40 seconds
  Interventions: Device: KXL System (45 mW/cm2); Drug: riboflavin ophthalmic solution

INTERVENTIONS:
Device: KXL System (15 mW/cm2) — UVA irradiation for 8 minutes at 15 mW/cm2
  Arms: VibeX Treatment Group A
Device: KXL System (30 mW/cm2) — UVA irradiation for 4 minutes at 30 mW/cm2
  Arms: VibeX Treatment Group B
Device: KXL System (45 mW/cm2) — UVA irradiation for 2 minutes 40 seconds at 45 mW/cm2
  Arms: VibeX Treatment Group C
Drug: riboflavin ophthalmic solution — Drops of riboflavin ophthalmic solution will be applied in the eye every two minutes for 20 minutes
  Other Names: VibeX

SUMMARY:
The objectives of this study are to evaluate and compare the safety and efficacy of three treatment regimens for corneal collagen cross-linking performed with VibeX (riboflavin ophthalmic solution) and the KXL System in impeding the progression of, and/or reducing maximum corneal curvature.

ELIGIBILITY:
Inclusion Criteria (all subjects):

1. Be at least 12 years of age, male or female, of any race;
2. Provide written informed consent and sign a HIPAA form. Patients who are under the age of 18 will need to sign an assent form as well as having a parent or legal guardian sign an informed consent;
3. Willingness and ability to follow all instructions and comply with schedule for follow-up visits;
4. For females capable of becoming pregnant, agree to have urine pregnancy testing performed prior to randomization of the study eye and on the day of the fellow eye treatment (which occurs between the 3 to 6 month study eye visits); must not be lactating, and must agree to use a medically acceptable form of birth control for at least one week prior to the randomization visit and continue to use the method until one month after the last dose of test article. Acceptable forms for birth control are spermicide with barrier, oral contraceptive, injectable or implantable method of contraception, transdermal contraceptive, intrauterine device, or surgical sterilization of partner. For non-sexually active females, abstinence will be considered an acceptable form of birth control. Women considered capable of becoming pregnant include all females who have experienced menarche and have not experienced menopause (as defined by amenorrhea for greater than 12 consecutive months) or have not undergone successful surgical sterilization (e.g. hysterectomy, bilateral tubal ligation, or bilateral oophorectomy);
5. BSCVA of ≥1 letter and ≤80 letters on ETDRS chart;
6. Presence of central or inferior steepening on the topographic map;
7. Contact Lens Wearers Only: Removal of contact lenses is required for a 1 week period prior to the screening visit(s);
8. Contact Lens Wearers Only: manifest refraction must be stable between two visits which occur at least 7 days apart. A stable refraction is one in which the manifest refraction spherical equivalent and the average K (Km) on the topographer taken at the first visit do not differ by more than 0.75 D from the respective measurements taken at the second exam;

   Inclusion Criteria (keratoconus subjects only):
9. Have a maximum corneal curvature as measured by Kmax of ≥ 47.00 D;
10. Having topographic evidence of keratoconus with a diagnosis of mild, moderate or severe keratoconus defined as the following:

    * Mild Keratoconus

      1. Axial topography consistent with keratoconus
      2. Flat keratometry reading ≤ 51.00 D on topography map
    * Moderate Keratoconus

      1. Axial topography consistent with keratoconus
      2. Flat keratometry reading ≥ 51.01 D and ≤ 56.00 D or astigmatism ≥ 8.00D on topography map
    * Severe Keratoconus:

      1. Axial topography consistent with keratoconus with marked areas of steepening
      2. Flat keratometry reading ≥ 56.01 D on topography map

    Inclusion Criteria (corneal ectasia subjects only):
11. Having a diagnosis of corneal ectasia after refractive surgery;
12. Having axial topography consistent with ectasia;

Exclusion Criteria (all subjects):

1. Contraindications, sensitivity or known allergy to the test article(s) or their components;
2. If female, be pregnant, nursing or planning a pregnancy or have a positive urine pregnancy test prior to the randomization or treatment of either eye or during the course of the study;
3. Corneal pachymetry that is < 375 microns prior to epithelial debridement at the thinnest point in the eye to be treated;
4. Eyes which are aphakic;
5. Eyes which are pseudophakic and do not have a UV blocking lens implanted;
6. Previous ocular condition (other than refractive error) in the eye to be treated that may predispose the eye for future complications. For example:

   1. History of corneal disease (e.g., herpes simplex, herpes zoster keratitis, recurrent erosion syndrome, corneal melt, corneal dystrophy, etc.)
   2. Clinically significant corneal scarring in the cross-linking treatment zone that is not related to keratoconus or corneal ectasia, in the investigator's opinion, will interfere with the cross-linking procedure;
7. A history of delayed epithelial healing in the eye(s) to be treated;
8. Patients with nystagmus or any other condition that would prevent a steady gaze during the treatment or other diagnostic tests;
9. Patients with a current condition that, in the investigator's opinion, would interfere with or prolong epithelial healing;
10. Taking Vitamin C (ascorbic acid) supplements within 1 week of the cross-linking treatment.
11. A history of previous corneal crosslinking treatment in the eye to be treated;
12. Have used an investigational drug or device within 30 days of the study or be concurrently enrolled in another investigational drug or device trial within 30 days of the study;
13. A history of previous corneal surgery (other than LASIK or PRK for subjects with corneal ectasia) or the insertion of Intacs in the eye(s) to be treated;
14. A history of previous Limbal Relaxing Incision (LRI) procedure in the eye(s) to be treated;
15. In addition, the Investigator may exclude or discontinue any subject for any sound medical reason;

    Exclusion Criteria (Keratoconus subjects only):
16. Eyes classified as either normal, atypical normal, or keratoconus suspect on the severity grading scheme.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1721 (Actual)
Dates: Start 2012-07; Primary Completion 2016-01 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Mean change in maximum corneal curvature (Kmax) from baseline | Month 6 or 12

SECONDARY OUTCOMES:
Comparison of treatment groups within each treatment indication | Month 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: John Vukich, MD, Principal Investigator — American-European Congress of Ophthalmic Surgery
Locations (83):
- United States (82):
  - John Parker, Birmingham, Alabama
  - Barnet Dulaney Perkins Eye Center, Phoenix, Arizona
  - Advanced Vision Care, Los Angeles, California
  - Stanford University School of Medicine, Palo Alto, California
  - Grutzmacher, Lewis and Sierra, Sacramento, California
  - Center for Sight, Sacramento, California
  - Newman Lasik Centers, Sacramento, California
  - Batra Vision Medical Group, San Leandro, California
  - Delta Eye Medical Group, Stockton, California
  - Kaiser Permanente - Kaiser Network Patients in Northern California Only, Walnut Creek, California
  - Mile High Corneal Specialists, PC, Denver, Colorado
  - Manchester Ophthalmology, Manchester, Connecticut
  - Eye Physicians and Surgeons, PC, Milford, Connecticut
  - TLC of Miami The Laser Center of Coral Gables, Coral Gables, Florida
  - Delray Eye Associates, PA, Delray Beach, Florida
  - Braverman Eye Center, Hallandale, Florida
  - The Eye Institute of West Florida, Largo, Florida
  - Herschel Lasik, Orlando, Florida
  - LCA-Vision Inc, Tampa, Florida
  - Quantum Vision Centers, Belleville, Illinois
  - University of Iowa Hospitals and Clinics, Coralville, Iowa
  - Kansas LasikPlus, P.A., Leawood, Kansas
  - Grene Vision Group, Wichita, Kansas
  - LaskiPlus Vision Center, Louisville, Kentucky
  - Ochsner Medical Center, New Orleans, Louisiana
  - Eyecare Medical Group, Portland, Maine
  - GBMC Dept. of Opthalmology/Mid-Atlantic Cornea Consultants, Baltimore, Maryland
  - Solomon Eye Physicians and Surgeons, Bowie, Maryland
  - Eye Doctors of Washington, Chevy Chase, Maryland
  - Boston Eye Group, Brookline, Massachusetts
  - Ophthalmic Consultants of Boston, Waltham, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Verdier Eye Center P.L.C., Grand Rapids, Michigan
  - Michigan Cornea Consultants, Southfield, Michigan
  - Chu Vision Institute, Bloomington, Minnesota
  - Eye Surgery and Laser Center, Madison, Mississippi
  - Pepose Vision Institute/ Lifelong Vision Foundation, Chesterfield, Missouri
  - Ophthamology Consultants LLC, St Louis, Missouri
  - The Eye Clinic Surgicenter, Billings, Montana
  - Eye Surgical Associates, Lincoln, Nebraska
  - Kugler Vision, PC, Omaha, Nebraska
  - Wellish Vision Institute, Las Vegas, Nevada
  - Princeton Eye Group, Princeton, New Jersey
  - Eye Associates of New Mexico, Albuquerque, New Mexico
  - CNY Eye Care, De Witt, New York
  - North Shore LIJ Health Systems, Great Neck, New York
  - Ramapo Ophthalmology Associates, LLP, Pomona, New York
  - Carolina Vision Center, Fayetteville, North Carolina
  - Bagan Strinden Vision, Fargo, North Dakota
  - Comprehensive Eye Care of Central Ohio, Westerville, Ohio
  - Dean McGee Eye Institute, Oklahoma City, Oklahoma
  - Devers Eye Institute, Portland, Oregon
  - Casey Eye Institute/OHSU, Portland, Oregon
  - Ophthalmic Partners of PA, P.C., Bala-Cynwyd, Pennsylvania
  - Schein Ernst Eye Associates, Harrisburg, Pennsylvania
  - Scheie Eye Institute, University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania
  - Corneal Associates, Wills Eye Institute, Philadelphia, Pennsylvania
  - Northeastern Eye Institute, Scranton, Pennsylvania
  - Bucci Laser Vision Institute, Wilkes-Barre, Pennsylvania
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Wright Vision Center, Rapid City, South Dakota
  - Vance Thompson Vision, Sioux Falls, South Dakota
  - Loden Vision Center, Goodlettsville, Tennessee
  - Wang Vision Institute, Nashville, Tennessee
  - Dell Laser Consultants, Austin, Texas
  - Buena Vista Eyecare, El Paso, Texas
  - Eye Consultants of Texas, Grapevine, Texas
  - Berkeley Eye Center, Houston, Texas
  - Slade and Baker Vision Center, Houston, Texas
  - Focal Point Vision, San Antonio, Texas
  - Hoopes Vision, Draper, Utah
  - The Eye Institute of Utah, Salt Lake City, Utah
  - University of Utah Dept. of Ophthalmology & Visual Sciences, Salt Lake City, Utah
  - Silk Vision & Surgical Center, Annandale, Virginia
  - Virginia Eye Consultants, Norfolk, Virginia
  - Commonwealth Eye Associates, Richmond, Virginia
  - Eye Care Center of Virginia, Richmond, Virginia
  - Beach Eye Care, Virginia Beach, Virginia
  - Evergreen Eye Center, Federal Way, Washington
  - Gundersen Clinic, Ltd., La Crosse, Wisconsin
  - Dean Foundation for Health, Research and Education, Inc., Madison, Wisconsin
- Lilia Rivera, San Juan, Puerto Rico